CLINICAL TRIAL: NCT05429853
Title: TOLER-ENT Study: A Study to Investigate the Tolerance of the High Energy, High Protein Formula Sondalis® HP 2 kcal
Acronym: SONDALIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been stopped prematurely for lack of inclusions
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-A03216-35
Record Dates: First submitted 2022-06-02; First posted 2022-06-23 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sondalis® HP 2 kcal (with or without fibre) (Experimental)
  Interventions: Dietary Supplement: Sondalis® HP 2 kcal (with or without fibre)

INTERVENTIONS:
Dietary Supplement: Sondalis® HP 2 kcal (with or without fibre) — The participants will take the study product during the two months of the study.

SUMMARY:
A multicentre, prospective, open-label, single arm study for 2 months, involving adult patients under poorly tolerated Home Enteral Nutrition (HEN). The study aims to analyse the evolution of tolerance and quality of life of HEN patients after switching from a High Protein High Energy (HPHE) polymeric Enteral Nutrition (EN) formula with or without fibre to Sondalis® HP 2kcal, with or without fibre. Eligible patients will give their written consent to participate before being included into the study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥18 years,
* Being under EN with polymeric HPHE product with or without fibre (=HPHE),
* Stable caloric prescription during HEN for at least one month,
* Patient with at least a score of 2 on at least 1 item of tolerance questionnaire,
* Investigators' judgement to change to HPHE concentrated,
* HEN is planned for ≥ 8 weeks,
* Life expectancy ≥ 3 months.
* Patient or his/her primary caregiver was required to be able to understand the study and to be fully free to participate in it,
* Patient having signed an informed consent,
* Patient registered with a social security scheme,
* Patient willing to adhere to study procedures,

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Being either under PN or ONS,
* Acute intestinal disease such as gastric ulcer, gastritis, gastroparesis,
* Patient under prokinetic agents during the study phase,
* Patient receiving antibiotic, chemotherapy in the 7 days prior to inclusion,
* Patient receiving radiation treatment except head and neck location,
* Patient expected to receive chemotherapy or radiation treatment during the study except head and neck location ,
* Severe infectious disease and/or fever > 38,5°C,
* Emergent hospitalization within last month,
* Known allergy or intolerance to any of the Sondalis® HP 2kcal with or without fibre ingredients,
* Previous treatment with HPHE concentrated at home (2kcal),
* Current participation in another intervention study or participation in a previous study for which exclusion period applies.
* Non-compliance with prescription and administration modalities as suspected by investigator and/or by home care provider dietitian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Evaluation tolerance from baseline after 2 months: Total Score | 60 days
  The digestive tolerance of enteral nutrition is assessed using a patient reported outcomes (PRO) questionnaire designed by clinicians. The questionnaire is composed of 9 items corresponding to the most frequent symptoms: gastro-oesophageal reflux, nausea, vomiting, feeling of an overfull stomach, bloating, flatulence, stomach pain, constipation, diarrhea. Each item includes questions relating to the frequency and impact of the symptom on daily life.

SECONDARY OUTCOMES:
Evaluation of Tolerance from baseline to one month and from one month to two months: Total Score | 60 days
  Same PRO than above
Evaluation of Tolerance at baseline,one and two months: for each Items | 60 days
  Same PRO than above
Evolution of quality of life | 60 days
  The quality of life is assessed with the NutriQoL® score described by Bischoff et al (Bischoff et al, 2020).
  The evolution of quality of life is evaluated between baseline, 1 month and 2 months after administration of the intervention.
  The NutriQoL® questionnaire is a specific tool to measure HRQoL in patients receiving HEN regardless of the underlying disease and the route of administration. It consists of 17 items grouped in two dimensions, which assess physical functioning, and activities of daily living and aspects of social life.
Evolution of anthropometric measures: handgrip test | 60 days
  The anthropometric measures are assessed with the handgrip test as recommended by SFNCM (Bossu-Estour et al, 2021).
  The evolution of anthropometric measures is evaluated between baseline, 1 month and 2 months after administration of the intervention.
  The Handgrip Test uses the Hand Grip Jamar® hydraulic hand dynamometers and the measurements are carried out according to the recommendations published by the "Comité Educationnel et de Pratique Clinique" of the SFNCM.
Evolution of anthropometric measures: body weight evolution | 60 days
  The anthropometric measures are assessed with the body weight evolution. The Weight is measured at the same time of day and under the same conditions (e.g. clothing).
Evolution of food intake | 30 days
  The food intake is assessed with the Food intake score (SEFI®). The evolution of food intake is evaluated between baseline, 1 month and 2 months after administration of the intervention.
  SEFI® allows a visual assessment of the patient's food intake, using a visual analogue scale, or a choice between consuming portions. The analogue scale is from 0: "I have eaten nothing" to 10: "I have eaten all".
Evolution of observance: score | 30 days
  The observance data are assessed with a score based on a questionnaire. The questionnaire assesses the frequency of difficulties in consuming the entire enteral nutrition prescription.
  The evolution of observance is evaluated between baseline, 1 month and 2 months after administration of the intervention.
Evolution of observance: number of bags | 30 days
  The observance data are assessed with the number of bags unused for 1 month. The evolution of observance is evaluated between baseline, 1 month and 2 months after administration of the intervention.
Evolution of Enteral Nutrition (EN) prescription procedure: Volume | 30 days
  The EN prescription procedure is assessed with the volume per 1 month administered.
  The evolution of EN prescription is evaluated between baseline, 1 month and 2 months after administration of the intervention.
Evolution of Enteral Nutrition (EN) prescription procedure: Time | 30 days
  The EN prescription procedure is assessed with the administration time per 1 month administered.
  The evolution of EN prescription is evaluated between baseline, 1 month and 2 months after administration of the intervention.
Evolution of Enteral Nutrition (EN) prescription procedure: Number of Bags | 30 days
  The EN prescription procedure is assessed with the number of bags per 1 month administered.
  The evolution of EN prescription is evaluated between baseline, 1 month and 2 months after administration of the intervention.
Evolution of Enteral Nutrition (EN) prescription procedure: Supplementary Hydration | 30 days
  The EN prescription procedure is assessed with the supplementary hydration per 1 month administered.
  The evolution of EN prescription is evaluated between baseline, 1 month and 2 months after administration of the intervention.
Safety events reporting | 60 days
  The safety is assessed with the report of safety events during the entire study period.
  Study adverse events are classified by system organ class (SOC), preferred terms (PT) in accordance with the current version of the Medical dictionary for Regulatory Activities (MedDRA), causality and seriousness.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane SCHNEIDER, Pr, Principal Investigator — Hôpital de l'Archet; David SEGUY, Pr, Principal Investigator — Hôpital Claude-Huriez
Locations (2):
- France (2):
  - Hôpital Claude Huriez, Lille
  - Hôpital de l'Archet, Nice